CLINICAL TRIAL: NCT04783623
Title: Analysis of Clinical Characteristics and Risk Factors of Recurrence of Endometriosis at Different Sites
Brief Title: Cohort Study of Endometriosis at Different Sites
Status: Completed | Type: Observational
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, XiaoyanLi, Primary investigator, Peking Union Medical College Hospital
Other Study IDs: S-K1522
Record Dates: First submitted 2021-03-02; First posted 2021-03-05 (Actual); Last update posted 2021-03-05 (Actual); Status verified 2021-03

CONDITIONS: Recruitment

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Non-recurrence group
  Interventions: Procedure: Surgical endometrioma excision
- Recurrence group
  Interventions: Procedure: Surgical endometrioma excision

INTERVENTIONS:
Procedure: Surgical endometrioma excision — We collect medical records of patients who had underwent surgical endometrioma excision at different sites in our hospital and conduct telephone or clinical interview

SUMMARY:
To present the clinical characteristics of pelvic or extra-pelvic endometriosis and explore the potential risk factors of pathogenesis and recurrence by comparing patients with endometriosis at different sites

DETAILED DESCRIPTION:
Endometriosis is a chronic inflammatory disease defined as the presence of endometrial glands and stroma outside of the internal epithelial lining of the cavum uteri, affecting up to 10% of reproductive age women. It is rarely found in extrapelvic locations.This form of endometriosis may be difficult to diagnosis due to pleomorphic presentation. Despite complete excision with a safe margin and histopathological examination has been considered as definitive diagnosis and primary therapeutic treatment for extra-pelvic endometriosis, what is understood mainly comes from case reports and retrospective observations with limited number of cases. Moreover, approximately 6%-14% of patients with PEM who had underwent narrowly operative resection still suffered recurrent lesions, while risk factors were barely identified.

Patients with endometriosis at different sites in our hospital were collected for analysis of clinical characteristics namely demographic information, medical history, surgical records, pathological and imaging reports, serum levels of cancer antigen 125 (CA125), peri-operative medication. During long-term follow-up, prognosis of individuals could be identified by telephone or clinical interview. Based on data from medical records or clinical observation, risk model predicting recurrence will be established by comparing patients with different outcomes or exposed to different risk factors. Thus, management of endometriosis might be improved. Hopefully, pathogenesis of recurrent and primary endometriosis might be explained.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were clinically diagnosed with endometriosis at different sites (pelvic and/or extra-pelvic) and received surgical treatment at PUMCH

Exclusion Criteria:

* i). underwent bilateral oophorectomy in the operation, ii). had incomplete records of inpatient management, iii). had no post-operative outpatient follow-up, iv). combined with malignancy.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women aged between 18 years old to 50 years old, who were diagnosed as endometriosis (both pelvic and extra-pelvic) and received surgical treatment in PUMCH.
Sampling Method: Non-Probability Sample
Enrollment: 146 (Actual)
Dates: Start 2021-01-20 (Actual); Primary Completion 2021-03-02 (Actual); Study Completion 2021-03-02 (Actual)

PRIMARY OUTCOMES:
clinicial outcome | 2 months
  recurrence or not

SECONDARY OUTCOMES:
clinical characteristics | 2 months
  Demographic information, medical history, surgical records, pathological and imaging reports (pelvic and/or trans-perineal and/or endorectal ultrasonography, computed tomography, magnetic resonance imaging), serum levels of cancer antigen 125 (CA125), perioperative medication

CONTACTS AND LOCATIONS:
Overall Officials: Jinhua Leng, Pro., Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No